CLINICAL TRIAL: NCT04976075
Title: Multicenter Prospective Observational and Epidemiological Registry for Patients With Intestinal Failure Due to Short Bowel Syndrome, in Latin America
Brief Title: ImpRovE underSTanding of Short bOwel syndRome in Latin-amErica
Acronym: RESTORE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: La Fundacion Favaloro para la Investigacion y la Docencia Medica (Other)
Collaborators: Fundación de Ciencias Exactas - UNLP (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Gabriel E. Gondolesi, Doctor, La Fundacion Favaloro para la Investigacion y la Docencia Medica
Other Study IDs: DDI 1384 1317 CBE 666-17
Record Dates: First submitted 2021-05-21; First posted 2021-07-26 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults: Patients of 18 or more years old
  Interventions: Other: no interventions
- Pediatrics: Patients less than 18 years old
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
Background and justification: Short bowel syndrome (SBS) is a disabling and life-threatening condition that results from a partial or total bowel resection, and has become as the main cause of Type III, intestinal failure (IF). Immediately after enterectomy there is an adaptation process consisting of structural, hormonal and metabolic changes to maximize intestinal function. These changes begin within days of resection and generally continue for several months. However, recent publications have reported even longer periods of time (up to 5 years) to achieve enteral autonomy.

It is possible to enhance the natural process of intestinal adaptation through medical or surgical treatments, called intestinal rehabilitation. During the process, complications related to intestinal failure or its treatment may arise, jeopardizing the result and even compromising survival. A better understanding of the medium and long-term results of patients under medical and / or surgical treatment with SIC is needed.

Despite the improvement recently achieved in managing IF, in most countries, pts are dispersed and seen by general health-care providers, with limited SBS or IF experience, causing increasing concern regarding the competence and equity of the care accessible to suffering pts.

The results obtained with the RESTORE project in adult patients highlight the relevance of having registries to better understand the natural history of this disease in adult patients, proving that a larger number of adult pts with SBS/III-IF can be identified and cared for than the numbers considered by recognized estimations. [Abstract sent to TTS, 2020].

To date, there are no data for pediatric patients with iIF secondary to SIC in Latin America, so its incidence, prevalence and evolution are unknown. Recent publications from middle-income countries, exposed the current inequality regarding the different types of therapies available within a given region.

Given the high morbidity and mortality associated with ICS-FI, there is an unmet need to create an adequate study that provides the information necessary to establish local and regional parameters and recommendations on its treatment.

DETAILED DESCRIPTION:
RESTORE amedment 1project, obtained the study number DDI (1384) 1317 from the Institutional Research and Ethics committee after its approving the choices of participating centers by RESTORE's Scientific Steering Committee. For participation, those centers needed a full-time or part-time surgeon-though not necessarily offing rehabilitation surgery or transplantation or accessing enterohormone (EH) therapies-a therapist with nutritional experience, a dietitian, and specialized pharmaceutical resources. Participating teams, however, did not necessarily have to offer rehabilitation surgery or transplantation capabilities or have access to EH therapies to be elected for participation.

RESTORE's aim was assessing the long-term outcomes of SBS pts with IF, under the current standard of care in order to plumb IF's natural history, the indications for currently available therapies, and their means of modifying each course.

Study Designed: the first prospective, observational, epidemiological, multicenter study in Argentina of adult pts with SBS-caused type-III IF in Lat-America.

In adults, the inclusion of additional centers in Argentina, Mexico, Colombia, Peru, Uruguay and Chile will be required. In pediatric patients, it is proposed to add patients and centers in Argentina and, if necessary, in other Latin American countries (Mexico, Colombia, Peru, Chile and Uruguay).

Number of patients and centers:

The study aims to recruit at least 150 patients in 24 centers. The sample size is based on the expected number of subjects who may be eligible and willing to participate in the study.

Diagnosis and inclusion criteria

Inclusion criteria:

1. Patients of both sexes, diagnosed with Type III-IF due to SBS
2. Signature of informed consent and assent as appropriate
3. 8 or more consecutive weeks of PN need

Exclusion criteria:

1. Less than 8 weeks of need for PN after diagnosis of SBS / IF
2. Refusal to provide informed consent and assent as appropriate
3. FI type I and II, and type III without SBS

The data from this study will be entered into an electronic CRF and database; with visits being reinitiated at weeks 4, 8, 12, 20, and 24 and then yearly thereafter. Pts that missed 2 or more visits were considered lost from follow-up. Death, recovery of intestinal sufficiency, and intestinal transplant were considered the end points.

The results of this study will be summarized and evaluated using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, diagnosed with Type III intestinal failure (FI) due to SIC
2. Signature of informed consent and assent as appropriate
3. 8 or more consecutive weeks of PN need

Exclusion Criteria:

1. Less than 8 weeks of need for PN after diagnosis of SIC / FI
2. Refusal to provide informed consent and assent as appropriate
3. FI type I and II, and type III without SIC

Ages: 1 Week to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Based on the SIC prevalence calculations, we aim to include 150 patients. The inclusion of patients will be done at the national level, considering as reference centers those hospitals that have Nutritional Support and Intestinal Rehabilitation Units, both public and private. Researchers may consecutively include all patients who give their consent and meet the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Describe the long term outcome of Type III-IF patients with short bowel syndrome in Latinoamérica. | April 2023
  The number of patients with short bowel syndrome/year, the number of patients able to recover intestinal sufficiency under the current available therapy that includes a) PN, b) medical and / or surgical rehabilitation, under the routine clinical practice in Latin American countries, will be reported. Long term survival (in months), freedom from Home Parenteral Nutrition survival in months, as measure for PN independence or recovery of intestinal insufficiency will be measured. The existence on post-surgical complications will be reported by using the Dindo-Clavien classification score (from 0 to 5).

SECONDARY OUTCOMES:
Describe the demographic characteristics and distribution of the disease | April 2023
  Type III-IF due to Short Bowel Syndrome patients' location will be descried.
Describe the nutritional progress | April 2023
  Nutritional progress (in Kgs and SGA) and growth (in cm, in children) in parallel with the assessment of the caloric intake (enteral and parenteral- in Kcal/week) and volume (l/week).
Record the use of Enterohormones | April 2023
  Those pts who could not continue decreasing HPN for 6-months, but had remained clinically stable, were considered candidates for EH therapies with the semisynthetic glucagon-like peptides 1 and 2 (sGLP-1, sGLP-2) according to each individual's need and potential benefit.
  In the sGLP-1 or sGLP-2 treatment, the initiation date, the clinical characteristics and course, and any adverse effects were recorded.
Describe the use, management of HPN, and its related complications | April 2023
  The HPN starting date, volume, kcals, and number of days per week were registered. HPN-related complications-including liver disease, catheter-related infections, central-venous-access loss, volume and/or caloric-requirement (kcal) changes throughout the course of care, or modifications in number of infusion days and volume during the treatment-were also registered and the ESPEN clinical classification recorded. Describe the incidence of PN-related complications: liver disease / failure associated with intestinal failure and PN, catheter-related infection, thrombosis, and loss of venous access.
Describe the surgical procedures, used, timing, outcomes and complications | April 2023
  Describe the surgical procedures used as part of intestinal rehabilitation, its complications and results CRATGI, or elongation surgery either with the Bianchi technique or STEP (Serial Transverse Enteroplasty). Postsurgical complications were registered after Dindo-Clavien's classification.
Assess the quality of life | April 2023
  Assess the quality of life (QoL) of patients under treatment (for the adult cohort) by using a brief survey assessing consistent in 3 questions to observe 3 main areas or domain: 1) Profesional/work performance, 2) Social activity and 3 Sexual Activity, based on a 0 to 10 index. Will be apply only o adult patients. .
Time to obtain therapy access | April 2023
  Time from from diagnoses to treatment access (in months) by age group and disease, will be asses.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Gondolesi, Doctor, Principal Investigator — University Hospital of the Favaloro Foundation
Locations (1):
- University Hospital of the Favaloro Foundation, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No